CLINICAL TRIAL: NCT01822600
Title: The Therapeutic Role of Albumin Supply on Peptic Ulcer Bleeding and the Correlation Between Clinical Course and Expression of Serum Response Factor on Ulcer Tissue and Superoxide Free Radical in Blood
Brief Title: The Therapeutic Role of Intravenous Albumin Administration for Peptic Ulcer Bleeding Patients With Hypoalbuminemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ER-98-239
Record Dates: First submitted 2013-03-20; First posted 2013-04-02 (Estimated); Last update posted 2019-08-29 (Actual); Status verified 2013-03

CONDITIONS: Peptic Ulcer Bleeding; Hypoalbuminemia
Keywords: hypoalbuminemia; peptic ulcer; rebleeding; hospitalization
MeSH Terms: conditions — Peptic Ulcer Hemorrhage; Hypoalbuminemia; Peptic Ulcer | interventions — Serum Albumin, Human; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Normal albumin group (Experimental): Based on the serum albumin level at enrollment, the patients were assigned into the normal albumin group if their serum albumin ≥ 30 g/L.
  Patients in this group receive intravenous omeprazole treatment.
  Interventions: Drug: Omeprazole
- Intervention group (Experimental): Based on the serum albumin level at enrollment, the patients were assigned into an intervention group if their serum albumin < 30 g/L.
  Patients in this group receive both Human albumin and intravenous omeprazole.
  Interventions: Drug: Human albumin; Drug: Omeprazole
- Cohort control group (Experimental): The study also included 29 patients with peptic ulcer bleeding and with hypoalbuminemia (serum albumin level < 30 g/L), but without receiving albumin supply from our previous study to serve as the cohort control group.
  Patients in this group receive intravenous omeprazole treatment.
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Human albumin — Each patient in the intervention group received Human Albumin 20%® (ZLB Behring, Marburg, Germany), immediately. The dosage of albumin infusion was 10 g q8h for 1 day in patients with albumin levels ranging from 25 g/L to 29 g/L or 2 days in those with albumin levels < 25 g/L.
  Other Names: Human Albumin 20%®, ZLB Behring, Marburg, Germany
  Arms: Intervention group
Drug: Omeprazole — After endoscopic hemostasis, each enrolled patient received an 80 mg loading dose of intravenous omeprazole (Losec®, AstraZeneca, Sweden) immediately. Patients then received a 3-day continuous omeprazole infusion in dosage of 80 mg per day.
  After omeprazole infusion, oral esomeprazole (Nexium®, AstraZeneca, Sweden) 40 mg per day was given in the normal albumin group and the intervention group until the end of follow-up.
  After omeprazole infusion, oral omeprazole (Losec®) 20 mg per day was given in the cohort control group until the end of follow-up.
  Other Names: Losec®, AstraZeneca, Sweden

SUMMARY:
To test whether intravenous albumin can decrease the rebleeding rate or shorten the duration of hospitalization in patients with peptic ulcer bleeding and hypoalbuminemia.

DETAILED DESCRIPTION:
Peptic ulcer bleeding is a common but potentially lethal disease. Recurrent bleeding is an independent risk factor for mortality. Inhibition of gastric acid secretion by intravenous proton pump inhibitor infusion can have a positive impact on the prevention of ulcer rebleeding after successful endoscopic therapy. However, the rebleeding rate can still be high in patients with comorbid illnesses even after proton pump inhibitor usage. Hypoalbuminemia has been reported to be a significant predictor of poor prognosis in patients with comorbid illnesses. Low serum albumin levels are associated with poor prognosis of wound healing and peptic ulcer bleeding; therefore, it is worthy to conduct a head-to-head comparison to validate whether administration of albumin can be helpful in improving the control of bleeding peptic ulcers, especially in patients with comorbid illnesses.

The albumin level may reflect upstream pathologic processes, such as stress or co-morbidities. Albumin administration may interrupt the downstream chain of poor outcome and thus maintain a favorable homeostasis in critically ill patients, and reduce morbidity. However, the clinical benefit of controlling peptic ulcer bleeding with exogenous albumin remains uncertain, and thus administration of albumin is not widely applied. Accordingly, the investigators conducted this pilot intervention to test whether short-term exogenous albumin administration can improve the control of peptic ulcer bleeding in hypoalbuminemic patients, who are at high risk of recurrent bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Clinical presentations of melena, hematochezia, or hematemesis
* Gastroscopy confirmed peptic ulcers and major stigmata of recent hemorrhage
* A Rockal score ≥ 6

Exclusion Criteria:

* Gastric or esophageal, or duodenal tumor bleeding
* Ulcer due to mechanical factors
* Warfarin use
* Failure to establish hemostasis under gastroscopy
* Hypersensitivity to omeprazole, esomeprazole, albumin or any component of the formulation.

Ages: 39 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2010-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
peptic ulcer rebleeding | within 28 days after the first bleeding event
  rebleeding was defined as: (i) continuous melena, hematochezia, or the presence of recurrent bloody aspirates through the naso-gastric tube; and (ii) relapse of hemodynamic instability, including systolic blood pressure < 90 mm Hg, heart rate >120 beats per min, or a hemoglobin drop by more than 20 g/L. For each patient with either suspected or active rebleeding of peptic ulcer, gastroscopy was conducted to confirm that the bleeding source was either a peptic ulcer or other non-ulcer conditions.

SECONDARY OUTCOMES:
the length of hospitalization | within 28 days after the first bleeding event
  the length of hospitalization after the first bleeding episode and the length of hospitalization after peptic ulcer rebleeding
the number of units of blood transfused | during the 28-day period after admission to the emergency room or after the presence of gastrointestinal bleeding signs in patients with nosocomial bleeding
the number of participants with massive rebleeding events in need of transarterial embolization or emergency surgery | within 28 days after the first bleeding event

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu-Chi Cheng, MD, PhD, Principal Investigator — Department of Internal Medicine, National Cheng Kung University Hospital, College of Medicine, National Cheng Kung University
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan